CLINICAL TRIAL: NCT03366857
Title: Effect of Supplemental Oxygen on Perioperative Brain Natriuretic Peptide Concentration in Cardiac Risk Patients - A Prospective Randomized Clinical Trial
Brief Title: Effect of Supplemental Oxygen on Perioperative BNP Concentration in Cardiac Risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Christian Reiterer, Dr. med. univ., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1744/2017
Record Dates: First submitted 2017-12-02; First posted 2017-12-08 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Supplemental Oxygen; Brain Natriuretic Peptide; Cardiac Risk Patients; Perioperative

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants don´t know the randomized oxygen concentration. The postoperative follow up will be performed by a blinded research fellow.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 30% (Active Comparator): Participants allocated to these groups will receive a FiO2 of 0.3 during the operation and for two hours postoperatively.
  Interventions: Drug: Oxygen 30 %
- 80% (Active Comparator): Participants allocated to these groups will receive a FiO2 of 0.8 during the operation and for two hours postoperatively.
  Interventions: Drug: Oxygen 80 %

INTERVENTIONS:
Drug: Oxygen 30 % — The oxygen concentration will be set at 30%.
  Arms: 30%
Drug: Oxygen 80 % — The oxygen concentration will be set at 80%.
  Arms: 80%

SUMMARY:
The effect of supplemental oxygen on surgical site infections was already investigated in several studies before. Although, oxygen is one of the most used medical therapy in hospitalized patients, the influence on the cardiovascular system is still unknown. Available data indicate beneficial effects of supplemental oxygen on cardiovascular function. Because, no evidence exists concerning the perioperative period, it is our objective to investigate supplemental oxygen in cardiac risk patients undergoing major abdominal surgery. Due to the significant reduction of BNP by inhibiting sympathetic nerve activity we hypothesize that supplemental oxygen have beneficial effects in perioperative BNP release in cardiac risk patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

Patients over 45 years on age, which fulfill 1 or more of the following 4 criteria undergoing non-cardiac surgery:

1. History of coronary artery disease
2. History of peripheral arterial disease
3. History of stroke OR
4. Any of 3 of 7 A) Age ≥ 70 years B) Undergoing major surgery C) History of congestive heart failure D) History of transient ischemic attack E) Diabetes and currently taking an oral hypoglycemic agent or insulin F) History of Hypertension

Further inclusion criteria are:

1. Written informed consent
2. Elective major abdominal open surgery or laparoscopically assisted procedures scheduled to take over two hours done under general anesthesia (colorectal, urology, gynecology, liver and pancreatic surgery)

Exclusion Criteria:

1. Symptoms of infection or sepsis
2. Preoperative inotropic therapy
3. Patients under ICU treatment
4. Oxygen dependent patients
5. History of severe heart failure and/or ejection fraction < 30%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Change of Postoperative Brain Natriuretic Peptide (BNP) concentration compared to preoperative baseline measurement during hospitalization | Preoperative, Postoperative (within 2 hours after end of surgery), Postoperative day 1 and 3 and within 72 hours before hospital discharge
  Perioperative BNP Concentration

SECONDARY OUTCOMES:
Redox Status - sORP (static oxidation-reduction potential), cORP (capacity oxidation-reduction potential) | Preoperative, 2 hours after induction of anesthesia, postoperative (within 2 hours after end of surgery), Postoperative day 1 and 3 and within 72 hours before hospital discharge
  Measurement of the Redox status using the RedoxSYS(R) system
Copeptin | Preoperative, Postoperative (within 2 hours after end of surgery), Postoperative day 1 and 3
  Perioperative plasma Copeptin concentration
MINS (myocardial ischemia after noncardiac surgery) | Preoperative, Postoperative (within 2 hours after end of surgery), Postoperative day 1 and 3
  Troponin T (TnT) measurement
vWF (von Willebrand factor) Antigen | Preoperative, Postoperative (within 2 hours after end of surgery), Postoperative day 1 and 3
  Effect of supplemental oxygen on inflammatory response using von Willebrand factor antigen
Fluid measurement | Intraoperative
  Due to the peripheral vasoconstriction of hyperoxia we measure the needed fluid for hemodynamic stability

CONTACTS AND LOCATIONS:
Overall Officials: Edith Fleischmann, Prof. Dr., Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria

REFERENCES:
- [Background] Meyhoff CS, Wetterslev J, Jorgensen LN, Henneberg SW, Hogdall C, Lundvall L, Svendsen PE, Mollerup H, Lunn TH, Simonsen I, Martinsen KR, Pulawska T, Bundgaard L, Bugge L, Hansen EG, Riber C, Gocht-Jensen P, Walker LR, Bendtsen A, Johansson G, Skovgaard N, Helto K, Poukinski A, Korshin A, Walli A, Bulut M, Carlsson PS, Rodt SA, Lundbech LB, Rask H, Buch N, Perdawid SK, Reza J, Jensen KV, Carlsen CG, Jensen FS, Rasmussen LS; PROXI Trial Group. Effect of high perioperative oxygen fraction on surgical site infection and pulmonary complications after abdominal surgery: the PROXI randomized clinical trial. JAMA. 2009 Oct 14;302(14):1543-50. doi: 10.1001/jama.2009.1452. PMID 19826023
- [Background] Greif R, Akca O, Horn EP, Kurz A, Sessler DI; Outcomes Research Group. Supplemental perioperative oxygen to reduce the incidence of surgical-wound infection. N Engl J Med. 2000 Jan 20;342(3):161-7. doi: 10.1056/NEJM200001203420303. PMID 10639541
- [Background] Shigemitsu M, Nishio K, Kusuyama T, Itoh S, Konno N, Katagiri T. Nocturnal oxygen therapy prevents progress of congestive heart failure with central sleep apnea. Int J Cardiol. 2007 Feb 14;115(3):354-60. doi: 10.1016/j.ijcard.2006.03.018. Epub 2006 Jun 23. PMID 16806535
- [Background] Rodseth RN, Biccard BM, Chu R, Lurati Buse GA, Thabane L, Bakhai A, Bolliger D, Cagini L, Cahill TJ, Cardinale D, Chong CP, Cnotliwy M, Di Somma S, Fahrner R, Lim WK, Mahla E, Le Manach Y, Manikandan R, Pyun WB, Rajagopalan S, Radovic M, Schutt RC, Sessler DI, Suttie S, Vanniyasingam T, Waliszek M, Devereaux PJ. Postoperative B-type natriuretic peptide for prediction of major cardiac events in patients undergoing noncardiac surgery: systematic review and individual patient meta-analysis. Anesthesiology. 2013 Aug;119(2):270-83. doi: 10.1097/ALN.0b013e31829083f1. PMID 23528538
- [Derived] Reiterer C, Fleischmann E, Kabon B, Taschner A, Kurz A, Adamowitsch N, von Sonnenburg MF, Fraunschiel M, Graf A. Hemodynamic effects of intraoperative 30% versus 80% oxygen concentrations: an exploratory analysis. Front Med (Lausanne). 2023 May 30;10:1200223. doi: 10.3389/fmed.2023.1200223. eCollection 2023. PMID 37324125
- [Derived] Reiterer C, Fleischmann E, Taschner A, Adamowitsch N, von Sonnenburg MF, Graf A, Fraunschiel M, Starlinger P, Goschin J, Kabon B. Perioperative supplemental oxygen and oxidative stress in patients undergoing moderate- to high-risk major abdominal surgery - A subanalysis of randomized clinical trial. J Clin Anesth. 2022 May;77:110614. doi: 10.1016/j.jclinane.2021.110614. Epub 2021 Nov 29. PMID 34856530
- [Derived] Reiterer C, Kabon B, Taschner A, Falkner von Sonnenburg M, Graf A, Adamowitsch N, Starlinger P, Goshin J, Fraunschiel M, Fleischmann E. Perioperative supplemental oxygen and NT-proBNP concentrations after major abdominal surgery - A prospective randomized clinical trial. J Clin Anesth. 2021 Oct;73:110379. doi: 10.1016/j.jclinane.2021.110379. Epub 2021 Jun 1. PMID 34087659
- [Derived] Reiterer C, Kabon B, von Sonnenburg MF, Starlinger P, Taschner A, Zotti O, Goshin J, Drlicek G, Fleischmann E. The effect of supplemental oxygen on perioperative brain natriuretic peptide concentration in cardiac risk patients - a protocol for a prosprective randomized clinical trial. Trials. 2020 May 12;21(1):400. doi: 10.1186/s13063-020-04336-9. PMID 32398119